CLINICAL TRIAL: NCT04794023
Title: A Combined First In Man And Pilot Study Investigating Visual And Refractive Outcomes In Lasik Surgery Using The Aquariuz Ablation Laser In Patients With Myopia, With Or Without Astigmatism
Brief Title: LASIK Surgery With a New Laser for the Treatment of Myopia Without Astigmatism
Acronym: AQUARIUZ2020
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ziemer Ophthalmic Systems AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZS004
Record Dates: First submitted 2021-03-04; First posted 2021-03-11 (Actual); Last update posted 2021-11-18 (Actual); Status verified 2021-04

CONDITIONS: Myopia; Astigmatism
Keywords: femtosecond LASIK; Solid state laser; AQUARIUZ; Corneal ablation
MeSH Terms: conditions — Myopia; Astigmatism

STUDY DESIGN:
Intervention Model Description: Phase I
  * Successful unilateral treatment of the dominant eye according to standard of care prior to investigational treatment
  * Unilateral investigational treatment on an amblyopic eye or a post-cataract eye
  * 4 eyes & 4 participants
  * Staged patient enrolment, to allow assessment and evaluation of safety parameters before investigational treatment is applied to the next participant
  * Interim analysis I - Verification of correction factor when all participants have reached 7 days follow-up
  Phase II
  * Initiated after Interim analysis I
  * Successful unilateral treatment of the dominant eye according to standard of care prior to investigational treatment
  * Unilateral investigational treatment on the non-dominant eye
  * 10 eyes & 10 participants
  * Interim analysis II - Confirmation of correction factor when all participants have reached 7 days follow-up
  Phase III
  * Initiated after Interim analysis II
  * Bilateral investigational treatment
  * 26 eyes & 13 participants
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention_Corneal Ablation (Experimental)
  Interventions: Device: Corneal Ablation

INTERVENTIONS:
Device: Corneal Ablation — Corneal ablation for the treatment of myopia with/without astigmatism following flap creation using femtosecond laser.

SUMMARY:
The AQUARIUZ ablation laser is a solid-state laser and has been CE approved for corneal surgery since March 2020 for the treatment of short- and longsightedness with and without astigmatism. The aim of this study is to collect the first clinical data. Safety and performance are examined here. The treatment with AQUARIUZ is comparable to treatments with an excimer laser, with the difference that these are operated with gas. Solid-state lasers and excimer lasers use the same process for tissue ablation, with a small difference in wavelength. This difference manifests itself in the lower involvement of water in the ablation process with the result of a gentler and safer treatment. Similar to excimer lasers for corneal surgery, the AQAURIUZ system (Ziemer Ophthalmic Systems AG) is equipped with a fast eye tracker (eye tracking system) to correct eye movements during the treatment. The shape of the removed portion of the cornea has an aspherical profile corresponding to the state of the art.

The primary objective is to assess the safety of use of the AQUARIUZ corneal ablation laser for LASIK procedures in myopia and myopia with astigmatism.

The secondary objective is to compare the predicted visual and refractive outcomes of LASIK procedures using the AQUARIUZ Ablation with clinical data.

The study is planned in 3 phases to mitigate the inherent risk of a first in man study and to allow for verification and confirmation of the system correction factor at an early stage.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria number 3 to 6, 10, 11 and 12 only apply to eyes planned for investigational treatment. Inclusion criterion number 9 applies to both eyes whether planned for investigational treatment or not and inclusion criterion number 8 applies to each eye as specified in the criteria.

  1. Informed Consent as documented by signature
  2. Medically suitable for corneal refractive surgery
  3. Stable refraction over a minimum of 12 months prior to surgery Stable refraction is defined as MRSE change per year in the eye to be treated ≤ 0.50 D and should be confirmed by at least one measurement between 1 and 10 years previous to the study.
  4. Myopia sphere from -0.5 D to -4.0 D
  5. Phases I & II: Maximum cylinder diopter -1.5 D
  6. Phase II & III: Maximum cylinder diopter -1.0 D
  7. Accurate baseline biometric measurements Accurate baseline biometric measurements are defined as

     * Assessed Manifest Refraction within ± 0.5 D of Objective Refraction
     * Less than 0.75 D spherical equivalent (SE) difference between cycloplegic and manifest refractions
     * Objective refraction should be assessed by

       * Autorefractometer And either/or
       * Hartmann-Shack Aberrometer
       * Ray tracing Aberrometer
  8. Age ≥ 18 years
  9. Calculated residual stroma thickness ≥ 300 microns
  10. IOP, as measured by non-contact tonometry < 21mmHg
  11. Phase I: One of the following

      * Amblyopic eye An amblyopic eye is defined as an eye that has decreased functional visual acuity due to an insufficient development in the visual system according to the judgement of the investigator, and the following criteria
      * Pre-operative CDVA up to 20/32 ( 0.63 in decimal convention)
      * Pre operative CDVA in the fellow, dominant eye ≥ 20/40 (0.5 in decimal convention)
      * Post-cataract patient, and the following criteria
      * Pre-operative CDVA in each eye ≥ 20/40 (0.5 in decimal convention)
  12. Phase II & III: Pre-operative CDVA in each eye ≥ 20/40 (0.5 in decimal convention)
  13. Patient willing and able to return to the study site for the follow-up visits, in the judgement of the investigator

Exclusion Criteria:

* The following exclusion criteria apply for both eyes, whether planned for treatment or not.

  1. Severe local infective or allergic conditions (e.g. blepharitis, past herpes simplex or zoster, allergic eye disease severe enough to require regular treatment).
  2. Corneal disease or pathology, such as but not limited to corneal scarring or opacity, history of viral keratitis, dry eye, recurrent epithelial erosion and Fuchs' endothelial dystrophy
  3. Manifest or subclinical keratoconus or keratectasia, as diagnosed by corneal topography and/or anterior optical coherence tomography
  4. Patients with degeneration of structures of the cornea, diagnosed keratoconus or any clinical pictures suggestive to keratoconus (form-fruste keratoconus)
  5. Corneal thickness < 480 microns
  6. Previous corneal surgery of any kind, including surgery for either refractive or therapeutic purposes in either eye that, in the judgement of the investigator confounds the outcome of the study or increases risk for the patient
  7. Glaucoma and/or ocular hypertension, whether untreated and under medical control
  8. Nystagmus or hemifacial spasm
  9. Known allergy to medications used in surgery, pre- and post-operative treatment at the investigational site
  10. Immunocompromised or diagnosis of ophthalmic disease (any of the following):

      * ocular herpes zoster or simplex
      * lupus
      * collagenases
      * other acute or chronic illnesses that increases the risk to the participant or confounds the outcomes of this study in the opinion of the investigator
  11. Patients with a diagnosed collagen vascular, atopic syndrome, autoimmune or immunodeficiency disease
  12. Known psychotic disorders associated with delusions (e.g. schizophrenia)
  13. Drug or alcohol abuse
  14. Neurological diagnosis with a GCS > 13
  15. Women who are pregnant or nursing or who plan to become pregnant over the course of this investigation.
  16. Inability to follow the procedures of the study in the opinion of the investigator, e.g. due to language problems, psychological disorders, dementia, etc.
  17. Participation in another interventional study within the 30 days preceding and during the present study
  18. Patients with uncontrolled diabetes
  19. Patients who are taking one or both of the following medications:

      * Isotretinoin (e.g. Accutane®)
      * Amiodarone hydrochloride (e.g. Cordarone®)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2021-03-31 (Actual); Primary Completion 2022-05 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Change between pre-operative CDVA and CDVA at 3 months follow-up | Baseline and 3 months
  Change between pre-operative CDVA and CDVA at 3 months follow-up:
  > 1 line loss from pre-operative CDVA
Number of unexpected Adverse Events | 3 months
  Unexpected adverse events (AEs) related to the device or the procedure under investigation, and that from the sponsor's or the principal investigator's point of view compromise patient safety
Number of Serious Adverse Events | 3 months
  SAEs related to the device or the procedure under investigation

SECONDARY OUTCOMES:
Change between pre-operative CDVA and post-operative UDVA | Baseline and 1-day
  The UDVA in decimal notation is defined as the inverse of the minimum angle of resolution (MAR) in a patients eye achieved without correction lenses or spectacles, measured over a distance of 4-6 metres by standardized letter charts .
  The CDVA is defined as the inverse of the minimum angle of resolution (MAR) in a patient's eye achieved with the best sphero-cylindrical prescription in trial lenses or spectacles, measured analogously to UDVA.
Change between pre-operative CDVA and post-operative UDVA | Baseline and 1 week
  The UDVA in decimal notation is defined as the inverse of the minimum angle of resolution (MAR) in a patients eye achieved without correction lenses or spectacles, measured over a distance of 4-6 metres by standardized letter charts .
  The CDVA is defined as the inverse of the minimum angle of resolution (MAR) in a patient's eye achieved with the best sphero-cylindrical prescription in trial lenses or spectacles, measured analogously to UDVA.
Change between pre-operative CDVA and post-operative UDVA | Baseline and 1 month
  The UDVA in decimal notation is defined as the inverse of the minimum angle of resolution (MAR) in a patients eye achieved without correction lenses or spectacles, measured over a distance of 4-6 metres by standardized letter charts .
  The CDVA is defined as the inverse of the minimum angle of resolution (MAR) in a patient's eye achieved with the best sphero-cylindrical prescription in trial lenses or spectacles, measured analogously to UDVA.
Change between pre-operative CDVA and post-operative UDVA | Baseline and 3 months
  The UDVA in decimal notation is defined as the inverse of the minimum angle of resolution (MAR) in a patients eye achieved without correction lenses or spectacles, measured over a distance of 4-6 metres by standardized letter charts .
  The CDVA is defined as the inverse of the minimum angle of resolution (MAR) in a patient's eye achieved with the best sphero-cylindrical prescription in trial lenses or spectacles, measured analogously to UDVA.
Change between pre-operative CDVA and post-operative UDVA | Baseline and 6 months
  The UDVA in decimal notation is defined as the inverse of the minimum angle of resolution (MAR) in a patients eye achieved without correction lenses or spectacles, measured over a distance of 4-6 metres by standardized letter charts .
  The CDVA is defined as the inverse of the minimum angle of resolution (MAR) in a patient's eye achieved with the best sphero-cylindrical prescription in trial lenses or spectacles, measured analogously to UDVA.
Change between pre-operative CDVA and post-operative UDVA | Baseline and 12 months
  The UDVA in decimal notation is defined as the inverse of the minimum angle of resolution (MAR) in a patients eye achieved without correction lenses or spectacles, measured over a distance of 4-6 metres by standardized letter charts .
  The CDVA is defined as the inverse of the minimum angle of resolution (MAR) in a patient's eye achieved with the best sphero-cylindrical prescription in trial lenses or spectacles, measured analogously to UDVA.
Difference between attempted versus achieved Manifest Refraction Spherical Equivalent (MRSE) after 1 week post surgery. | Baseline and 1 week
  The MRSE is defined as the mean refractive deficit in diopters (D) over two main meridians as assessed by monocular sphero-cylindrical refraction (manifest refraction).
  The manifest refraction is a set of three numerical, continues variables (Spherical dioptres - MRSPH, cylindrical dioptres - MRCYL, cylindrical axis in degrees).
  MRSE is deduced from the manifest refraction as follows:
  MRSE = MRSPH + ½ x MRCYL
Difference between attempted versus achieved Manifest Refraction Spherical Equivalent (MRSE) after 1 month post surgery. | Baseline and 1 month
  The MRSE is defined as the mean refractive deficit in diopters (D) over two main meridians as assessed by monocular sphero-cylindrical refraction (manifest refraction).
  The manifest refraction is a set of three numerical, continues variables (Spherical dioptres - MRSPH, cylindrical dioptres - MRCYL, cylindrical axis in degrees).
  MRSE is deduced from the manifest refraction as follows:
  MRSE = MRSPH + ½ x MRCYL
Difference between attempted versus achieved Manifest Refraction Spherical Equivalent (MRSE) after 3 months post surgery. | Baseline and 3 months
  The MRSE is defined as the mean refractive deficit in diopters (D) over two main meridians as assessed by monocular sphero-cylindrical refraction (manifest refraction).
  The manifest refraction is a set of three numerical, continues variables (Spherical dioptres - MRSPH, cylindrical dioptres - MRCYL, cylindrical axis in degrees).
  MRSE is deduced from the manifest refraction as follows:
  MRSE = MRSPH + ½ x MRCYL
Difference between attempted versus achieved Manifest Refraction Spherical Equivalent (MRSE) after 6 months post surgery. | Baseline and 6 months
  The MRSE is defined as the mean refractive deficit in diopters (D) over two main meridians as assessed by monocular sphero-cylindrical refraction (manifest refraction).
  The manifest refraction is a set of three numerical, continues variables (Spherical dioptres - MRSPH, cylindrical dioptres - MRCYL, cylindrical axis in degrees).
  MRSE is deduced from the manifest refraction as follows:
  MRSE = MRSPH + ½ x MRCYL
Difference between attempted versus achieved Manifest Refraction Spherical Equivalent (MRSE) after 12 months post surgery. | Baseline and 12 months
  The MRSE is defined as the mean refractive deficit in diopters (D) over two main meridians as assessed by monocular sphero-cylindrical refraction (manifest refraction).
  The manifest refraction is a set of three numerical, continues variables (Spherical dioptres - MRSPH, cylindrical dioptres - MRCYL, cylindrical axis in degrees).
  MRSE is deduced from the manifest refraction as follows:
  MRSE = MRSPH + ½ x MRCYL
Percentage of eyes within ±0.5 D, and ±1 D of the attempted MRSE after 1 week post surgery. | Baseline and 1 week
Percentage of eyes within ±0.5 D, and ±1 D of the attempted MRSE after 1 month post surgery. | Baseline and 1 month
Percentage of eyes within ±0.5 D, and ±1 D of the attempted MRSE after 3 months post surgery. | Baseline and 3 months
Percentage of eyes within ±0.5 D, and ±1 D of the attempted MRSE after 6 months post surgery. | Baseline and 6 months
Percentage of eyes within ±0.5 D, and ±1 D of the attempted MRSE after 12 months post surgery. | Baseline and 12 months
Observed difference in manifest refraction after 1 week post surgery. | Baseline and 1 week
  The manifest refraction is a set of three numerical continues variables (Spherical dioptres - MRSPH, cylindrical dioptres - MRCYL, cylindrical axis in degrees).
Observed difference in manifest refraction after 1 month post surgery. | Baseline and 1 month
  The manifest refraction is a set of three numerical continues variables (Spherical dioptres - MRSPH, cylindrical dioptres - MRCYL, cylindrical axis in degrees).
Observed difference in manifest refraction after 3 months post surgery. | Baseline and 3 months
  The manifest refraction is a set of three numerical continues variables (Spherical dioptres - MRSPH, cylindrical dioptres - MRCYL, cylindrical axis in degrees).
Observed difference in manifest refraction after 6 months post surgery. | Baseline and 6 months
  The manifest refraction is a set of three numerical continues variables (Spherical dioptres - MRSPH, cylindrical dioptres - MRCYL, cylindrical axis in degrees).
Observed difference in manifest refraction after 12 months post surgery. | Baseline and 12 months
  The manifest refraction is a set of three numerical continues variables (Spherical dioptres - MRSPH, cylindrical dioptres - MRCYL, cylindrical axis in degrees).
Difference (in terms of cylindrical power and orientation of meridians) between Target Induced Astigmatism (TIA) versus Surgically Induced Astigmatism (SIA) after 1 week post surgery. | Baseline and 1 week
Difference (in terms of cylindrical power and orientation of meridians) between pre-operative and post-operative magnitude of astigmatism after 1 month post surgery. | Baseline and 1 month
Difference (in terms of cylindrical power and orientation of meridians) between pre-operative and post-operative magnitude of astigmatism after 3 months post surgery. | Baseline and 3 months
Difference (in terms of cylindrical power and orientation of meridians) between pre-operative and post-operative magnitude of astigmatism after 6 months post surgery. | Baseline and 6 months
Difference (in terms of cylindrical power and orientation of meridians) between pre-operative and post-operative magnitude of astigmatism after 12 months post surgery. | Baseline and 12 months
Angle of error, defined as the angle described by the vectors of the achieved correction (SIA) versus the intended correction (TIA) after 1 week post surgery. | Baseline and 1 week
  The angle of error is positive if the achieved correction is on an axis counterclockwise (CCW) to where it was intended and negative if the achieved correction is clockwise (CW) to its intended axis.
  The astigmatism vector is the combination of the magnitude, MRCYL, and the cylindrical axis in degrees and will be assessed as described above. Vector analysis will be performed according to Alpins et al 2001 and Thibos et al 2001.
Angle of error, defined as the angle described by the vectors of the achieved correction (SIA) versus the intended correction (TIA) after 1 month post surgery. | Baseline and 1 month
  The angle of error is positive if the achieved correction is on an axis counterclockwise (CCW) to where it was intended and negative if the achieved correction is clockwise (CW) to its intended axis.
  The astigmatism vector is the combination of the magnitude, MRCYL, and the cylindrical axis in degrees and will be assessed as described above. Vector analysis will be performed according to Alpins et al 2001 and Thibos et al 2001.
Angle of error, defined as the angle described by the vectors of the achieved correction (SIA) versus the intended correction (TIA) after 3 months post surgery. | Baseline and 3 months
  The angle of error is positive if the achieved correction is on an axis counterclockwise (CCW) to where it was intended and negative if the achieved correction is clockwise (CW) to its intended axis.
  The astigmatism vector is the combination of the magnitude, MRCYL, and the cylindrical axis in degrees and will be assessed as described above. Vector analysis will be performed according to Alpins et al 2001 and Thibos et al 2001.
Angle of error, defined as the angle described by the vectors of the achieved correction (SIA) versus the intended correction (TIA) after 6 months post surgery. | Baseline and 6 months
  The angle of error is positive if the achieved correction is on an axis counterclockwise (CCW) to where it was intended and negative if the achieved correction is clockwise (CW) to its intended axis.
  The astigmatism vector is the combination of the magnitude, MRCYL, and the cylindrical axis in degrees and will be assessed as described above. Vector analysis will be performed according to Alpins et al 2001 and Thibos et al 2001.
Angle of error, defined as the angle described by the vectors of the achieved correction (SIA) versus the intended correction (TIA) after 12 months post surgery. | Baseline and 12 months
  The angle of error is positive if the achieved correction is on an axis counterclockwise (CCW) to where it was intended and negative if the achieved correction is clockwise (CW) to its intended axis.
  The astigmatism vector is the combination of the magnitude, MRCYL, and the cylindrical axis in degrees and will be assessed as described above. Vector analysis will be performed according to Alpins et al 2001 and Thibos et al 2001.

OTHER OUTCOMES:
Change between pre-operative CDVA and CDVA after 1 week post surgery. | Baseline and 1 week
Change between pre-operative CDVA and CDVA after 1 month post surgery. | Baseline and 1 month
Change between pre-operative CDVA and CDVA after 6 months post surgery. | Baseline and 6 months
Change between pre-operative CDVA and CDVA after 12 months post surgery. | Baseline and 12 months
Number of unexpected Adverse Events after 1 week post surgery. | 1 week
  Unexpected adverse events (AEs) related to the device or the procedure under investigation, and that from the sponsor's or the principal investigator's point of view compromise patient safety
Number of unexpected Adverse Events after 1 month post surgery. | 1 month
  Unexpected adverse events (AEs) related to the device or the procedure under investigation, and that from the sponsor's or the principal investigator's point of view compromise patient safety
Number of unexpected Adverse Events after 6 months post surgery. | 6 months
  Unexpected adverse events (AEs) related to the device or the procedure under investigation, and that from the sponsor's or the principal investigator's point of view compromise patient safety
Number of unexpected Adverse Events after 12 months post surgery. | 12 months
  Unexpected adverse events (AEs) related to the device or the procedure under investigation, and that from the sponsor's or the principal investigator's point of view compromise patient safety
Number of Serious Adverse Events after 1 week post surgery. | 1 week
  SAEs related to the device or the procedure under investigation
Number of Serious Adverse Events after 1 month post surgery. | 1 month
  SAEs related to the device or the procedure under investigation
Number of Serious Adverse Events after 6 months post surgery. | 6 months
  SAEs related to the device or the procedure under investigation
Number of Serious Adverse Events after 12 months post surgery. | 12 months
  SAEs related to the device or the procedure under investigation

CONTACTS AND LOCATIONS:
Locations (1):
- Augen Glattzentrum ONO Wallisellen, Wallisellen, Canton Zürich, Switzerland